CLINICAL TRIAL: NCT00094757
Title: A Multicenter, Randomized, Double-Blind Study of MK0431 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: An Investigational Drug Study in Patients With Type 2 Diabetes Mellitus (MK0431-023)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-023; 2004_045
Record Dates: First submitted 2004-10-22; First posted 2004-10-25 (Estimated); Results first posted 2010-07-21 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Sitagliptin 100 mg (Experimental): Sitagliptin 100 mg
  Interventions: Drug: Comparator: sitagliptin 100 mg
- Sitagliptin 200 mg (Experimental): Sitagliptin 200 mg
  Interventions: Drug: Comparator: sitagliptin 200 mg
- Placebo/Pioglitazone (Placebo Comparator): Placebo/Pioglitazone
  Interventions: Drug: Comparator: placebo; Drug: Comparator: pioglitazone

INTERVENTIONS:
Drug: Comparator: sitagliptin 100 mg — sitagliptin 100 mg oral tablet once daily for 54 weeks
  Arms: Sitagliptin 100 mg
Drug: Comparator: sitagliptin 200 mg — sitagliptin 200 mg (2- 100 mg oral tablets) once daily for 54 weeks
  Arms: Sitagliptin 200 mg
Drug: Comparator: placebo — placebo oral tablet once daily during Phase A (Weeks 0-18)
  Arms: Placebo/Pioglitazone
Drug: Comparator: pioglitazone — pioglitazone 30 mg oral tablet once daily during Phase B (Weeks 18-54)
  Arms: Placebo/Pioglitazone

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an investigational drug in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age and not older than 75 who have a specific type of diabetes called Type 2 Diabetes Mellitus

Exclusion Criteria:

* Younger than 18 years of age or older than 75
* Any condition, which in the opinion of the investigator, may not be in the patient's best interest to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2004-10-06 (Actual); Primary Completion 2005-08-17 (Actual); Study Completion 2006-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Raz I, Hanefeld M, Xu L, Caria C, Williams-Herman D, Khatami H; Sitagliptin Study 023 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor sitagliptin as monotherapy in patients with type 2 diabetes mellitus. Diabetologia. 2006 Nov;49(11):2564-71. doi: 10.1007/s00125-006-0416-z. Epub 2006 Sep 26. PMID 17001471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 15-Oct-2004. Last Patient Last Visit: 28-Apr-2006. 60 medical clinics in the United States (US), 37 in 4 countries in Europe, and 17 in 5 countries in the rest of the world.
Pre-assignment Details: Patients 18-75 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control (Hemoglobin A1C ≥7% and ≤10.0%) on diet and exercise alone were eligible to enter the study.
Groups:
- Sitagliptin 100 mg: The Sitagliptin 100 mg got 1 sitagliptin 100 mg tablet and 1 sitagliptin matching placebo tablet once daily Weeks 0-54 and pioglitazone placebo once daily in Weeks 18-54.
- Sitagliptin 200 mg: The Sitagliptin 200 mg got 2 sitagliptin 100 mg tablets once daily Weeks 0-54 and pioglitazone placebo once daily in Weeks 18-54.
- Placebo/Pioglitazone: The Placebo/Pioglitazone got 2 sitagliptin matching placebo tablets once daily in Weeks 0- 54 and pioglitazone 30 mg/day once daily in Weeks 18-54.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Started | 205 | 206 | 110
Completed | 152 | 144 | 80
Not Completed | 53 | 62 | 30
Not completed — Adverse Event | 11 | 9 | 6
Not completed — Lack of Efficacy | 11 | 15 | 8
Not completed — Lost to Follow-up | 3 | 5 | 6
Not completed — Patient Moved | 2 | 1 | 1
Not completed — Protocol Violation | 8 | 5 | 3
Not completed — Withdrawal by Subject | 14 | 21 | 5
Not completed — Other | 3 | 3 | 1
Not completed — Protocol specified discontinuation | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone | Total
Number analyzed (Participants) | 205 | 206 | 110 | 521
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.0) | 55.4 (9.2) | 55.5 (10.1) | 55.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 102 | 41 | 238
  Male | 110 | 104 | 69 | 283
Race/Ethnicity, Customized [Number; unit: participants]
  White | 142 | 146 | 68 | 356
  Black | 16 | 11 | 12 | 39
  Hispanic | 37 | 39 | 22 | 98
  Asian | 8 | 7 | 5 | 20
  Other | 2 | 3 | 3 | 8
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent] | 8.0 (0.8) | 8.1 (0.9) | 8.0 (0.9) | 8.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 18
Description: Hemoglobin A1C (A1C) is measured as percent. Thus this change from baseline reflects the Week 18 A1C percent minus the Week 0 A1C percent.
Time Frame: Weeks 0-18
Population: All Patients Treated included those with ≥1 dose of study therapy, had a baseline and ≥1 post-baseline value. For those with no data at Week 18, last post-baseline observation was carried forward. Data after initiation of glycemic rescue were considered missing. Analysis adjusted for baseline values and prior antihyperglycemic therapy status.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Number analyzed (Participants) | 193 | 199 | 103
percent | -0.48 [-0.61 to -0.35] | -0.36 [-0.48 to -0.23] | 0.12 [-0.05 to 0.30]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo/Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA — Model terms: treatment, baseline, prior anti-hyperglycemic therapy status (on vs. not on prior therapy); Mean Difference (Net) = -0.60, 95% CI 2-sided [-0.82 to -0.39], Standard Deviation 0.90
Statistical Analysis 2: Comparison: Sitagliptin 200 mg vs Placebo/Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline, prior anti-hyperglycemic therapy status (on vs. not on prior therapy); Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.70 to -0.26], Standard Deviation 0.90

2. Secondary Outcome: Change From Baseline in FPG at Week 18
Description: The change from baseline reflects the Week 18 Fasting Plasma Glucose (FPG) minus the Week 0 FPG.
Time Frame: Weeks 0-18
Population: All Patients Treated included patients who received at least 1 dose of study therapy, and had a baseline value and ≥1 post-baseline value for this outcome. The last post-baseline observed measurement was carried forward to Week 18 for patients with no data at Week 18. Data after initiation of glycemic rescue were considered missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Number analyzed (Participants) | 201 | 202 | 107
mg/dL | -12.7 [-19.1 to -6.3] | -9.9 [-16.2 to -3.5] | 7.0 [-1.8 to 15.8]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo/Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline, prior anti-hyperglycemic therapy status; Mean Difference (Net) = -19.7, 95% CI 2-sided [-30.5 to -8.9], Standard Deviation 45.9
Statistical Analysis 2: Comparison: Sitagliptin 200 mg vs Placebo/Pioglitazone; Test type: Superiority or Other; p < 0.002, ANCOVA; Model terms: treatment, baseline, prior anti-hyperglycemic therapy status; Mean Difference (Net) = -16.9, 95% CI 2-sided [-27.6 to -6.1], Standard Deviation 45.9

3. Secondary Outcome: Change From Baseline in A1C at Week 54
Description: A1C is measured as percent. Thus this change from baseline reflects the Week 54 A1C percent minus the Week 0 A1C percent.
Time Frame: Weeks 0-54
Population: All Patients Treated included patients who received at least 1 dose of study therapy post-Week 18, a baseline value and ≥1 post-Week 18 value for this outcome. The last post- Week 18 observed measurement was carried forward to Week 54 for patients with no data at Week 54. Data after initiation of glycemic rescue were considered missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Number analyzed (Participants) | 156 | 158 | 68
percent | -0.28 [-0.42 to -0.14] | -0.19 [-0.33 to -0.05] | -0.87 [-1.08 to -0.66]

4. Secondary Outcome: Change From Baseline in FPG at Week 54
Description: The change from baseline reflects the Week 54 FPG minus the Week 0 FPG.
Time Frame: Weeks 0-54
Population: All Patients Treated included patients who received at least 1 dose of study therapy 1 post-Week 18, a baseline value and ≥1 post-Week 18 value for this outcome. The last post- Week 18 observed measurement was carried forward to Week 54 for patients with no data at Week 54. Data after initiation of glycemic rescue were considered missing.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Number analyzed (Participants) | 159 | 160 | 70
mg/dL | -5.5 [-11.5 to 0.5] | -0.7 [-6.7 to 5.3] | -28.0 [-37.1 to -18.9]

ADVERSE EVENTS:
Time Frame: Weeks 0 to 54
Description: Patients received rescue medication if they met specific glycemic goals. SAEs include events that occurred either before or after receiving rescue medication. Other AEs only includes those AEs that occurred prior to a patient receiving rescue medication.
Arm/Group | Sitagliptin 100 mg | Sitagliptin 200 mg | Placebo/Pioglitazone
Serious Adverse Events (participants affected / at risk) | 15/205 | 12/206 | 10/110
Other Adverse Events (participants affected / at risk) | 70/205 | 55/206 | 37/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=205) | Sitagliptin 200 mg (N=206) | Placebo/Pioglitazone (N=110)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1
Complication Of Device Insertion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Polytraumatism (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood Potassium Decreased (Investigations) | 0 | 1 | 0
Blood Sodium Decreased (Investigations) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0 | 0
Bladder Perforation (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Leriche Syndrome (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 100 mg (N=205) | Sitagliptin 200 mg (N=206) | Placebo/Pioglitazone (N=110)
Influenza (Infections and infestations) | 11 | 8 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 14 | 6
Urinary Tract Infection (Infections and infestations) | 8 | 10 | 9
Blood Glucose Increased (Investigations) | 17 | 7 | 9
Glycosylated Haemoglobin Increased (Investigations) | 11 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 11 | 5
Headache (Nervous system disorders) | 13 | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.